CLINICAL TRIAL: NCT00010881
Title: Oregon Center for Complementary and Alternative Medicine in Neurological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Purpose: Treatment
Other Study IDs: P50 AT000066-01M; P50AT000066-01 (NIH); NCT00009451 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Neurological Disorders
MeSH Terms: conditions — Nervous System Diseases | interventions — Antioxidants; Mindfulness-Based Stress Reduction

INTERVENTIONS:
Drug: antioxidants
Behavioral: stress reduction

SUMMARY:
The mission of the Oregon Center for Complementary and Alternative Medicine in Neurological Disorders (ORCCAMIND) is to facilitate research and education on the effectiveness and mechanisms of action of complementary and alternative medicine (CAM) therapies in the treatment of neurological disorders. The integration of conventional medicine and CAM communities is critical for the success of ORCCAMIND. Thus, ORCCAMIND is composed of six institutions: Oregon Health Sciences University; National College of Naturopathic Medicine; Western States Chiropractic College; Oregon College of Oriental Medicine; the Linus Pauling Institute at Oregon State University; and the Portland Veterans Affairs Medical Center.

ORCCAMIND will initially focus on the use of CAM antioxidants and stress reduction as treatments for neurodegenerative and demyelinating diseases because many of these diseases have oxidative injury as a causative or contributory factor and several CAM approaches have direct or indirect anti-oxidant effects. Through the Career Development Program the Developmental Research Program and the activities of the Education and Information Core, we will also foster and promote research into other CAM approaches for neurologic diseases that extend beyond anti-oxidant therapies. ORCCAMIND will achieve its goals by carrying out 4 Research Projects and maintaining 4 Core facilities that integrate the research strengths of conventional medicine and CAM practitioners and researchers. ORCCAMIND draws its strength from the multi-institutional support and the quality of all its investigators. The investigators join ORCCCAMIND with extensive experience with clinical trials, patient care, externally funded basic and clinical neuroscience research, and training programs, including federally-funded training grants. ORCCAMIND is a bold initiative that integrates basic and clinical research scientists, conventional neurologists and CAM practitioners. It will promote the exploration of new areas of CAM research and lead research on CAM therapies for neurological disorders.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* written informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 1999-09; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Barry S. Oken, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health Sciences Univ./Neurology, Portland, Oregon, United States